CLINICAL TRIAL: NCT02679456
Title: A Multicenter, Randomized, Evaluator Blinded, Active-Controlled Study to Evaluate the Safety and Efficacy of Oral Ibrexafungerp (SCY-078) vs. Oral Fluconazole in Subjects With Vulvovaginal Candidiasis
Brief Title: Safety and Efficacy of Oral Ibrexafungerp (SCY-078) vs. Oral Fluconazole in Subjects With Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCY-078-203
Record Dates: First submitted 2016-01-19; First posted 2016-02-10 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — ibrexafungerp; Fluconazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group 1 (Fluconazole) (Active Comparator): Fluconazole
  Interventions: Drug: Fluconazole
- Treatment Group 2: (SCY-078) (Experimental): Dose regimen 1
  Interventions: Drug: SCY-078
- Treatment Group 3 (SCY-078) (Experimental): Dose regimen 2
  Interventions: Drug: SCY-078

INTERVENTIONS:
Drug: SCY-078
  Arms: Treatment Group 2: (SCY-078); Treatment Group 3 (SCY-078)
Drug: Fluconazole
  Arms: Treatment Group 1 (Fluconazole)

SUMMARY:
This is a randomized, multicenter, evaluator blinded study to evaluate the safety, tolerability, efficacy and pharmacokinetics of SCY-078 compared to Fluconazole in adult patients with moderate to severe Vulvovaginal Candidiasis (VVC) and a history of frequent episodes of VVC. Approximately 90 subjects, meeting the inclusion criteria will be enrolled and randomized in a 1:1:1 ratio to one of the 3 treatment arms: Oral SCY-078 in 2 dose regimens or oral Fluconazole. After enrollment, subjects will be evaluated on Day-5 (end of treatment visit), Day-24 (test of cure visit), Day-60, Day 90 and Day 120 (end of observation period visit) or at any time that a recurrence or clinical failure is suspected, up to the end of observation period.

DETAILED DESCRIPTION:
This is a randomized, multicenter, evaluator blinded study to evaluate the safety, tolerability, efficacy and pharmacokinetics of SCY-078 compared to Fluconazole in adult patients, from 18 to 65 years of age, with moderate to severe Vulvovaginal Candidiasis (VVC) and a history of frequent episodes of VVC. Approximately 90 subjects, meeting the inclusion criteria will be enrolled and randomized in a 1:1:1 ratio to one of the 3 treatment arms: oral SCY-078 does regimen 1, or oral SCY-078 does regimen 2, or oral Fluconazole. After enrollment, subjects will be evaluated on Day-5 (end of treatment visit), Day-24 (test of cure visit), Day-60, Day 90 and Day 120 (end of observation period visit) or at any time that a recurrence or clinical failure is suspected, up to the end of observation period.

Primary Objectives:

* To evaluate the safety and efficacy of 2 dosing regimens of Oral SCY-078 in subjects with moderate to severe Vulvovaginal Candidiasis (VVC)

Secondary Objectives:

* To estimate the effect of Oral SCY-078 therapy in the rate and time to recurrence in subjects with a history of frequent episodes of VVC

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be eligible for study admission:

1. Female subjects from 18 to 65 years of age in good general health
2. Diagnosis of symptomatic moderate to severe vulvovaginal candidiasis
3. The ability to understand and sign a written informed consent form (ICF), which must be obtained prior to treatment and any study-related procedures.
4. The ability to understand and sign a consent or authorization form which shall permit the use, disclosure and transfer of the subject's personal health information (e.g., in the U.S. HIPAA Authorization form).
5. The ability to understand and follow all study-related procedures including study drug administration.
6. Females of childbearing potential must agree to use a medically acceptable method of contraception while receiving protocol-assigned product.

Exclusion Criteria:

A subject will be excluded from participation in the study if she meets any of the following exclusion criteria:

1. Any vaginal condition other than VVC that may interfere with the diagnosis or evaluation of response to therapy.
2. Prior use of any prohibited medication(s) or procedure(s) within the protocol specified timeframe including:

   a. Systemic and/or topical (vaginal) antifungal treatment, prescription or over the counter, within 30 days of the baseline visit.
3. Subjects with history of renal impairment, hepatic impairment or cervical cancer.

4 Subjects with known hypersensitivity to enfumafungin derivatives, fluconazole or any of the components of the formulation.

5. HIV infection, chemotherapy or illness serious enough to induce an immune deficiency.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving therapeutic cure at the test of cure visit (Day 24 +/-3) | Day 24 +/- 3
  Therapeutic Cure defined as achieving both a Clinical Cure (resolution of signs and symptoms) and a Mycological Eradication (negative culture).

SECONDARY OUTCOMES:
Proportion of subjects with recurrence of VVC during the observation period | 4-month observation period
  Recurrence defined as a symptomatic and culture-verified episode of VVC after achieving Therapeutic Cure.

CONTACTS AND LOCATIONS:
Overall Officials: David Angulo, MD, Study Director — Scynexis, Inc.
Locations (2):
- Dominican Republic (2):
  - Hospital Dr. Francisco E. Moscoso Puello, Santo Domingo
  - Instituto Dermatologico y Cirugia de Piel, Santo Domingo

IPD SHARING:
Plan to Share IPD: Undecided